CLINICAL TRIAL: NCT03276468
Title: A Phase II Trial Evaluating Combination of Atezolizumab, With Venetoclax and Obinutuzumab for Relapsed/Refractory Lymphomas
Brief Title: Evaluation of Atezolizumab-Venetoclax-Obinutuzumab Combination in Relapse/Refractory Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GATA
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Follicular Lymphoma; Diffuse Large B Cell Lymphoma; Marginal Zone Lymphoma; Mucosa Associated Lymphoid Tissue
Keywords: venetoclax; obinutuzumab; atezolizumab; lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone; Lymphoma | interventions — atezolizumab; obinutuzumab; venetoclax

STUDY DESIGN:
Intervention Model Description: This study is a multicentric open-label phase II trial in 3 cohorts of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Combination of venetoclax, atezolizumab and obinutuzumab
  Interventions: Drug: Atezolizumab; Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg on day 2 of each 21-day cycle during 18 months (24 cycles)
  Other Names: Tecentriq
Drug: Obinutuzumab — 1000 mg on day 1, day 8 and day 15 of cycle 1 and each day 1 from cycle 2 to cycle 8
  Other Names: Gazyvaro
Drug: Venetoclax — 800 mg/d from day 8 of cycle 1, every day during 18 months. For MZL patients wiht lymphocytes>5 g/l : 50 mg/day: week 1 100mg/day: week 2 200mg/day: week 3 400mg/day: week 4 800mg/day: from week 5
  Other Names: Venclyxto

SUMMARY:
This study is a multicenter phase II trial which primary objective is to assess the anti-lymphoma activity of atezolizumab associated with a BCL-2 inhibitor (GDC-199, venetoclax) and an anti-CD20 monoclonal antibody (obinutuzumab) in three separate cohorts:

* relapsed/refractory follicular lymphoma (FL) patients
* relapsed/refractory aggressive (DLBCL) lymphoma patients
* relapsed/refractory other indolent (iNHL) lymphoma patients (MZL and MALT)

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented CD20-positive follicular lymphoma (WHO grade 1, 2, or 3a) patients for cohort 1
* Patients with either histologically documented CD20-positive Diffuse large-cell lymphoma (including transformations of low-grade lymphoma into DLBCL) or follicular lymphoma CD20+ grade 3b, or primary cutaneous DLBCL leg type, or primary mediastinal (thymic) large B-cell lymphoma, or high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, or unclassifiable B-cell lymphoma with features intermediate between DLBCL and Hodgkin (WHO classification) for cohort 2
* Patients with relapsed/refractory indolent lymphoma (marginal zone (MZL) or measurable mucosa-associated lymphoid tissue (MALT) lymphoma) for cohort 3
* Relapsed/refractory NHL after ≥1 prior R-containing regimen with no curative option
* Aged 18 years or more with no upper age limit
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Bi-dimensionally measurable disease defined by at least one single node or tumor lesion > 1.5 cm assessed by CT scan, or Positron Emission Tomography (PET) scan without IV contrast at diagnosis with at least one hypermetabolic lesion
* Signed written informed consent
* Life expectancy ≥ 3 months
* Females of childbearing potential (FCBP) must agree to use one reliable form of contraception or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 18 months after discontinuation of all study treatments
* Male patients and their partner (FCBP) must agree to use two reliable forms of contraception (condom for males and hormonal method for partners) during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 18 months after discontinuation of all study treatments
* Patient covered by any social security system

Exclusion Criteria:

* Lymphocytic lymphoma (LL), waldenström macroglobulinemia, unmeasurable MALT lymphoma, Mantle Cell Lymphoma (MCL) and Follicular lymphoma for cohort 3
* Known CD20 negative status at last biopsy done (Biopsy at relapse/progression is mandatory)
* Central nervous system or meningeal involvement by lymphoma
* Prior history of Progressive Multifocal Leukoencephalopathy (PML)
* Documented infection with HIV
* Active Hepatitis B (HB) (positive Hepatitis B surface antigen (Ag-HBs) OR positive serology to hepatitis B (positive Ag-HBs or Hepatitis B core antibody (anti-HBc) or Polymerisation Chain Reaction (PCR) for viral DNA of HBV) Active Hepatitis C (HC) infection (patients with positive HCV serology (anti-HCV) are eligible only if PCR is negative from known HCV RNA)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) before inclusion, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to first administration of study drug
* Active immune-related disease criteria
* Left Ventricular Ejection Fraction (LVEF) < 45% as determined by echocardiography or multiple uptake gated acquisition (MUGA) scan
* Any serious active disease or co-morbid medical condition (such as New York Heart Association Class III or IV cardiac disease, severe arrhythmia, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including uncontrolled obstructive pulmonary disease and history of bronchospasm or other according to investigator's decision)
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Any of the following laboratory abnormalities:
* Hemoglobin < 9 g/dL
* Absolute neutrophil count (ANC) < 1,000 cells/mm3 (1.0 G/L) unless due to lymphoma
* Platelet count < 75,000/mm3 (75 x 109/L) unless due to lymphoma
* Serum glutamic-oxaloacetic transaminase (SGOT) / Aspartate Transaminase (AST) or Serum Glutamic-Pyruvate Transferase (SGPT) / Alanine Transaminase (ALT) 3.0 x upper limit of normal (ULN) unless disease involvement
* Serum total bilirubin > 2.0 mg/dL (34 μmol/L), except if disease related or in case of Gilbert syndrome
* Calculated creatinine clearance (Cockcroft-Gault formula or MDRD) of < 50 mL /min
* International normalized ratio (INR) ≤ 1.5 x ULN for patients not receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) or activated PTT (aPTT) > 1.5 x ULN
* Prior history of malignancies other than lymphoma unless the subject has been free of the disease for ≥ 3 years. Exceptions will be allowed for patients with non-melanoma skin tumors (basal cell or squamous cell carcinoma of the skin) or any surgically removed stage 0 (in situ) carcinoma
* Any serious medical condition, laboratory abnormality (other than mentioned above), or psychiatric illness that would prevent the subject from signing the informed consent form
* Contraindication to any drug contained in the study treatment regimen
* Previous treatment with obinutuzumab, atezolizumab or venetoclax
* Use of any standard or experimental anti-cancer drug therapy within 28 days prior to first administration of study drug
* Use of warfarin prior to first administration of study drug and throughout all treatment period (because of potential drug-drug interactions that may potentially increase the exposure of warfarin)
* Patients taking corticosteroids within 4 weeks prior to first administration of study drug, unless administered at a cumulated dose equivalent to ≤ 3.5mg/kg (within these 4 weeks).
* Use of the following agents prior to first administration of study drug: Strong and moderate CYP3A inhibitors (including grapefruit juice); Strong and moderate CYP3A inducers
* Pregnant or lactating females
* Person deprived of his/her liberty by a judicial or administrative decision
* Adult person under legal protection
* Person hospitalized without consent
* Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
FL and DLBCL cohorts : Overall Metabolic Response Rate (OMRR) at the end of induction | 8 months (8 cycles)
  Assessment of disease response according to Lugano 2014
for iNHL cohort : Overall Response Rate (ORR) at the end of induction | 8 months (8 cycles)
  Assessment of disease response according to Lugano 2014

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 4 years
  time from inclusion to the first observation of progression
Overall Survival (OS) | 4 years
  time from inclusion to death
Duration of Response (DR) | 4 years
  from a confirmed Complete Metabolic Response / Complete Radiologic Response (CMR/CRR) or Partial Metabolic Response / Partial Radiologic Response (PMR/PRR) the first observation of progression
for FL and DLBCL cohorts : OMRR | 4 months, 18 months
  According to Lugano 2014
for iNHL cohort : ORR | 4 months, 18 months
  According to Lugano 2014
Best response | 18 months
  Percentage of each response type according to Lugano 2014

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CARTRON, PhD, Principal Investigator — Lymphoma Study Association; Charles HERBAUX, MD, Principal Investigator — Lymphoma Study Association
Locations (25):
- France (25):
  - CHU d'Angers, Angers
  - CHU de Caen, Caen
  - CHU de Clermont Ferrand - Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CH Annecy Gennevois, Épagny
  - CHD de Vendée, La Roche-sur-Yon
  - CHU de Grenoble, La Tronche
  - CHRU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy - Brabois, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Necker, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU de Rennes - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - CHRU de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No